CLINICAL TRIAL: NCT02486835
Title: Efficacy & Tolerability of a Specific Plantain,Thyme and Honey Cough Syrup vs Placebo in Child Cough Due to Common Cold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Avner Herman Cohen, Prof. Herman Avner Cohen, Clalit Health Services
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABO-cough-2015
Record Dates: First submitted 2015-05-17; First posted 2015-07-01 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Cough Syrup for adults and children" (Experimental): Marked (authorized) medical device acting by protecting the oropharynx, in a non pharmacological way, to reduce cough. It contains honey, plantago lanceolata, thymus vulgaris.Dosage form: syrup Dosage: 5 ml three times a day. Frequency: the duration of the study for each patient is 4 nights, 3 days.
  Interventions: Device: Cough syrup for adults and children
- Placebo (Placebo Comparator): The placebo intervention is a syrup of same taste and colour without the protective components. Dosage form: syrup. Dosage: 5 ml three times a day Frequency: the duration of the study for each patient is 4 nights, 3 days.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Cough syrup for adults and children — Dosage is 5 ml three times a day for 4 nights, 3 days
  Other Names: Poliflav M.A.-honey cough syrup
  Arms: "Cough Syrup for adults and children"
Device: Placebo — Dosage is 5 ml three times a day for 4 nights, 3 days
  Arms: Placebo

SUMMARY:
Cough is a life saving reflex, therefore it is important, especially in pediatrics, to calm cough spells without sedating the reflex. The intent of this study is to use a protective syrup with does not act as a sedative or as a potent mucolytic and measure its efficacy and safety versus placebo in children with moderate to severe night and daily cough. Cough is assessed with a validated parent questionnaire. The degree of disturbance of cough is followed immediately after one night administration of the study products and daily for 4 nights, 3 days.

DETAILED DESCRIPTION:
Cough is a life saving reflex, therefore it is important, especially in pediatrics, to calm cough spells without sedating the reflex. Looking into mechanisms for cough management different from mucolytics, or sedatives, such as protection of irritated pharynx mucosa from post nasal drip or other irritating substances is theoretically sound and shows practical interesting results.

A parallel comparison of efficacy and tolerability between such protective mechanism (acting through a barrier and radical scavenging action) due to natural substances (honey, plantago lanceolata and thymus vulgaris) and placebo has not been done so far, in very young children, especially in a time frame of 4 days. The intent of this study is to use the protective syrup versus placebo in children with moderate to severe night and daily cough, measured with a validated parent questionnaire. The degree of disturbance of cough is followed immediately after one night administration of the study products and daily for 4 nights, 3 days.

Assessment of effectiveness of the protective cough syrup as compared to placebo is considered very interesting due to the mechanism of the remedy.

ELIGIBILITY:
Inclusion Criteria:

* cough attributed to infection of the upper respiratory tract since less or equal than 7 days,
* children aged 1 to 5 years
* score of three or more of al least two of the following three questions relating to night cough, frequency of nocturnal cough, impact on sleep of child and impact on sleep of parent,
* score of at least three of all questions assessing daytime cough considering the day prior to study entry
* written consent by a parent.

Exclusion Criteria:

* Children with a diagnosis of acute laryngotracheal bronchitis, pneumonia, asthma, sinusitis, allergic rhinitis, as well as chronic cardiac condition, or cystic fibrosis or any anatomical respiratory tract anomalies,
* Children who received antihistamines or any cough medicine the day prior to study entry,
* The administration of any steroid preparation by oral administration or inhalation on the day prior to study entry,
* Known sensitivity to any component of placebo or to Plantago lanceolata or Thymus vulgaris, honey or any other component of the cough syrup.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2016-04-03 (Actual); Study Completion 2016-04-06 (Actual)

PRIMARY OUTCOMES:
Change in night cough frequency score in the general population | baseline up to night 1
  Night cough frequency is the most invasive element of distress to the child and family. The questionnaire rating night cough is filled in each morning relating to the passed night for four nights. The basal night score is the score of the night before enrollment.

SECONDARY OUTCOMES:
Change in night cough frequency score in the population coughing since 1-2 days | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in night cough frequency score in the female population coughing since 1-2 days | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in night cough frequency score in the male population coughing since 1-2 days | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in night cough severity score in the general population | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in night cough severity score in the population coughing since 1-2 days | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in night cough bothersomeness score in the general population | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in night cough bothersomeness score in the population coughing since 1-2 days | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in night cough influence on sleep of child score in the general population | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in night cough influence on sleep of child score in the population coughing since 1-2 days | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in night cough influence on sleep of parent score in the general population | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in night cough influence on sleep of parent score in the population coughing since 1-2 days | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in night cough combined score in the general population | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in night cough combined score in the population coughing since 1-2 days | baseline up to night 1
  All these other elements constitute cough invasiveness into the quality of life of child and parents
Change in day cough frequency score in the general population | baseline up to day 2
  The questionnaire rating day cough is filled in each evening relating to the passed day for three days.
  The basal day score is the score of the day before enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Herman A Cohen, Prof., Principal Investigator — Clalit HS
Locations (4):
- Israel (4):
  - Pediatric Ambulatory Clinic Bat-Yam, Bat Yam
  - Pediatric Ambulatory Clinic Kfar-Saba, Kfar Saba
  - Pediatric Community Ambulatory Clinic - Petach-Tikva, Petah Tikva
  - Pediatric Ambulatory Clinic Ramat Aviv Gimel, Tel Aviv

REFERENCES:
- [Background] Middleton KR, Hing E. National Hospital Ambulatory Medical Care Survey: 2004 outpatient department summary. Adv Data. 2006 Jun 23;(373):1-27. PMID 16841784
- [Background] Paul IM, Yoder KE, Crowell KR, Shaffer ML, McMillan HS, Carlson LC, Dilworth DA, Berlin CM Jr. Effect of dextromethorphan, diphenhydramine, and placebo on nocturnal cough and sleep quality for coughing children and their parents. Pediatrics. 2004 Jul;114(1):e85-90. doi: 10.1542/peds.114.1.e85. PMID 15231978
- [Background] Paul IM, Beiler J, McMonagle A, Shaffer ML, Duda L, Berlin CM Jr. Effect of honey, dextromethorphan, and no treatment on nocturnal cough and sleep quality for coughing children and their parents. Arch Pediatr Adolesc Med. 2007 Dec;161(12):1140-6. doi: 10.1001/archpedi.161.12.1140. PMID 18056558
- [Background] Wegener T, Kraft K. [Plantain (Plantago lanceolata L.): anti-inflammatory action in upper respiratory tract infections]. Wien Med Wochenschr. 1999;149(8-10):211-6. German. PMID 10483683
- [Background] Canciani M, Murgia V, Caimmi D, Anapurapu S, Licari A, Marseglia GL. Efficacy of Grintuss(R) pediatric syrup in treating cough in children: a randomized, multicenter, double blind, placebo-controlled clinical trial. Ital J Pediatr. 2014 Jun 10;40:56. doi: 10.1186/1824-7288-40-56. PMID 24917119
- [Background] Rimsza ME, Newberry S. Unexpected infant deaths associated with use of cough and cold medications. Pediatrics. 2008 Aug;122(2):e318-22. doi: 10.1542/peds.2007-3813. PMID 18676517
- [Background] Schramm DD, Karim M, Schrader HR, Holt RR, Cardetti M, Keen CL. Honey with high levels of antioxidants can provide protection to healthy human subjects. J Agric Food Chem. 2003 Mar 12;51(6):1732-5. doi: 10.1021/jf025928k. PMID 12617614
- [Background] Bogdanov S, Jurendic T, Sieber R, Gallmann P. Honey for nutrition and health: a review. J Am Coll Nutr. 2008 Dec;27(6):677-89. doi: 10.1080/07315724.2008.10719745. PMID 19155427
- [Background] Cohen HA, Rozen J, Kristal H, Laks Y, Berkovitch M, Uziel Y, Kozer E, Pomeranz A, Efrat H. Effect of honey on nocturnal cough and sleep quality: a double-blind, randomized, placebo-controlled study. Pediatrics. 2012 Sep;130(3):465-71. doi: 10.1542/peds.2011-3075. Epub 2012 Aug 6. PMID 22869830